CLINICAL TRIAL: NCT02106676
Title: Androgen Metabolism and Reproductive Outcome
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 03
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Polycystic Ovary Syndrome; Healthy Pregnant Women
Keywords: polycystic ovary Syndrome; hyperandrogenism; cordblood; androgens
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant women with PCOS and offspring: Exposures of interest: Polycystic ovary Syndrome (PCOS) according to Rotterdam
- Pregnant women without PCOS and offspring: Exposures of interest: Pregnant women without polycystic ovary Syndrome (PCOS) according to Rotterdam

SUMMARY:
The aim of this study is to determine maternal androgen metabolism during pregnancy and the impact of androgen disorders on mothers and infants.

DETAILED DESCRIPTION:
Women with polycystic ovary syndrome (PCOS) have an impaired fertility and significant higher complication rates during infertility treatment, pregnancy and the perinatal period. Complications include the occurrence of multiple gestations, ovarian hyper stimulation syndrome, early pregnancy loss, gestational diabetes, pregnancy-induced hypertension, pre-eclampsia and need for caesarean section. Moreover, their infants are more frequently born preterm, have higher perinatal mortality rates and are more often admitted to a neonatal intensive care unit. The etiology of PCOS is not particularly mapped, but a genetic background can be assumed by analyzing PCOS families. In utero androgen excess has also been suspected to be an important risk factor. Animal studies have demonstrated that intrauterine hyperandrogenic environment affects the offspring by leading to biochemical and morphological features of PCOS. Sex differences in prenatal androgen levels have been observed and testosterone levels in umbilical cord blood and in amniotic fluid are higher in healthy male babies than in healthy female babies. There are just a few reporting on the relation between maternal androgen levels during pregnancy and the respective offspring. The aim of this clinical study is to determine maternal androgen metabolism and the impact of androgen disorders on mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with and without PCOS

Exclusion Criteria:

* unable to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Polycystic ovary Syndrome (PCOS): According to ethnicity and the criteria used for diagnosis, polycystic ovary syndrome (PCOS) affects between 2-13% of women of reproductive age (Asunción et al., 2000; Azziz et al., 2009; ESHRE/ASRM, 2004; Wang and Alvero, 2013).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
correlation of testosterone between mother and offspring | day of birth (within average 24 hours)

SECONDARY OUTCOMES:
correlation of sexual hormon binding globulin between mother and offspring | day of birth (within average 24 hours)
correlation of thyroid-stimulating hormone between mother and offspring | day of birth (within average 24 hours)
correlation of androstendione between mother and offspring | day of birth (within average 24 hours)
correlation of anti muellerian hormon between mother and offspring | day of birth (within average 24 hours)
correlation of progesterone between mother and offspring | day of birth (within average 24 hours)
correlation of dehydroepiandrosteron between mother and offspring | day of birth (within average 24 hours)
correlation of Vitamin D levels between mother and offspring | day of birth (within average 24 hours)
correlation of prolactin between mother and offspring | day of birth (within average 24 hours)
correlation of insulin between mother and offspring | day of birth (within average 24 hours)
correlation of human growth hormon between mother and offspring | day of birth (within average 24 hours)
correlation of c-peptide between mother and offspring | day of birth (within average 24 hours)
correlation of cortisol between mother and offspring | day of birth (within average 24 hours)
correlation of luteinizing hormon between mother and offspring | day of birth (within average 24 hours)
correlation of follicle stimulating hormone between mother and offspring | day of birth (within average 24 hours)
correlation of estrogen levels between mother and offspring | day of birth (within average 24 hours)
maternal testosterone | six weeks after birth
maternal sexual hormon binding globulin | six weeks after birth
maternal thyroid-stimulating hormone | six weeks after birth
maternal androstendione | six weeks after birth
maternal anti muellerian hormon | six weeks after birth
maternal progesterone | six weeks after birth
maternal dehydroepiandrosteron | six weeks after birth
maternal Vitamin D levels | six weeks after birth
maternal prolactin | six weeks after birth
maternal insulin | six weeks after birth
maternal human growth hormon | six weeks after birth
maternal c-peptide | six weeks after birth
maternal cortisol | six weeks after birth
maternal luteinizing hormon | six weeks after birth
maternal follicle stimulating hormone | six weeks after birth
maternal estrogen levels | six weeks after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Background] Barry JA, Kay AR, Navaratnarajah R, Iqbal S, Bamfo JE, David AL, Hines M, Hardiman PJ. Umbilical vein testosterone in female infants born to mothers with polycystic ovary syndrome is elevated to male levels. J Obstet Gynaecol. 2010;30(5):444-6. doi: 10.3109/01443615.2010.485254. PMID 20604643
- [Background] Anderson H, Fogel N, Grebe SK, Singh RJ, Taylor RL, Dunaif A. Infants of women with polycystic ovary syndrome have lower cord blood androstenedione and estradiol levels. J Clin Endocrinol Metab. 2010 May;95(5):2180-6. doi: 10.1210/jc.2009-2651. Epub 2010 Mar 12. PMID 20228162
- [Background] Abbott DH, Barnett DK, Bruns CM, Dumesic DA. Androgen excess fetal programming of female reproduction: a developmental aetiology for polycystic ovary syndrome? Hum Reprod Update. 2005 Jul-Aug;11(4):357-74. doi: 10.1093/humupd/dmi013. PMID 15941725
- [Background] van de Beek C, Thijssen JH, Cohen-Kettenis PT, van Goozen SH, Buitelaar JK. Relationships between sex hormones assessed in amniotic fluid, and maternal and umbilical cord serum: what is the best source of information to investigate the effects of fetal hormonal exposure? Horm Behav. 2004 Dec;46(5):663-9. doi: 10.1016/j.yhbeh.2004.06.010. PMID 15555509
- [Background] Hickey M, Sloboda DM, Atkinson HC, Doherty DA, Franks S, Norman RJ, Newnham JP, Hart R. The relationship between maternal and umbilical cord androgen levels and polycystic ovary syndrome in adolescence: a prospective cohort study. J Clin Endocrinol Metab. 2009 Oct;94(10):3714-20. doi: 10.1210/jc.2009-0544. Epub 2009 Jun 30. PMID 19567524
- [Background] Norman RJ, Dewailly D, Legro RS, Hickey TE. Polycystic ovary syndrome. Lancet. 2007 Aug 25;370(9588):685-97. doi: 10.1016/S0140-6736(07)61345-2. PMID 17720020
- [Background] Goodarzi MO, Guo X, Yildiz BO, Stanczyk FZ, Azziz R. Correlation of adrenocorticotropin steroid levels between women with polycystic ovary syndrome and their sisters. Am J Obstet Gynecol. 2007 Apr;196(4):398.e1-5; discussion 398.e5-6. doi: 10.1016/j.ajog.2006.12.009. PMID 17403434